CLINICAL TRIAL: NCT00376506
Title: A Comparison of an Implanted Neuroprosthesis With Sensory Training for Improving Airway Protection in Chronic Dysphagia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 060212; 06-N-0212
Record Dates: First submitted 2006-09-14; First posted 2006-09-15 (Estimated); Results first posted 2012-10-26 (Estimated); Last update posted 2012-10-26 (Estimated); Status verified 2012-09

CONDITIONS: Chronic Dysphagia; Multiple Sclerosis; Parkinson Disease
Keywords: Aspiration; Rehabilitation; Swallowing Disorders; Stroke; Parkinson's Disease; Dysphagia; Parkinson Disease; PD
MeSH Terms: conditions — Multiple Sclerosis; Parkinson Disease; Deglutition Disorders; Stroke

ARMS (2):
- Implanted Device (Experimental): Implanted intramuscular neurostimulator device
  Interventions: Device: Neurostimulation device for dysphagia
- External Device (Active Comparator): External vibrotactile device
  Interventions: Device: External vibrotactile device

INTERVENTIONS:
Device: Neurostimulation device for dysphagia — A neurostimulation device that is surgically implanted in the swallowing muscles.
  Arms: Implanted Device
Device: External vibrotactile device — A vibrotactile device that is placed on the neck during swallowing.
  Arms: External Device

SUMMARY:
This study will compare an implant with the technique of sensory training to determine which method may improve the ability to swallow and reduce the risk of choking. Many people with a brain injury or neurological disorders experience difficulty in swallowing. Past studies have shown that an electrical pulse applied to muscles or an increase in sensory stimulation to the throat can help.

Patients ages 18 to 90 who have had a brain injury or neurological disorder and who have had trouble swallowing for 6 months or longer may be eligible for this study. Patients will undergo a physical examination, pregnancy test, and exam by a throat and speech physician. Fiber-optic endoscopic evaluation of swallowing with sensory testing involves a flexible tube passed through the nose to the back of the throat to allow observation of the voice box. Videofluoroscopy, an X-ray of the head and neck, will be done while patients swallow. Patients experiencing trouble with the upper esophagus may undergo additional procedures, including manometry to measure pressure changes in the back of the throat, and reevaluation through the fiber-optic tube. Patients in this study will have a magnetic resonance imaging (MRI) scan, which uses a strong magnetic field to obtain images of the body. Patients will lie on a table that slides into the enclosed tunnel of the scanner. The scan will take 20 to 25 minutes.

Patients will be assigned randomly to one of two groups: the intramuscular group, to have a stimulation device implanted in the neck, and the vibrotactile group, to receive a vibrotactile stimulator. All patients will have 10 training sessions with their devices, plus follow-up. Those patients in the first group will undergo surgery, under general anesthesia, for the implant. Three weeks following the implant procedure, patients will come to NIH to have the stimulator turned on and programmed and to learn how to use the device. Those patients in the second group will have about 2 to 3 weeks of training in using a vibrotactile device, and then they will take it home to use. All patients will return to NIH at 3 months to ensure proper use of the devices, and they will visit for follow-up at 6 months and 12 months for tests and questionnaires.

...

DETAILED DESCRIPTION:
Objective: To determine if an implanted neuroprosthesis improves airway protection for swallowing in chronic pharyngeal dysphagia to a greater degree than sensory training. The implanted neuroprosthesis will provide intramuscular stimulation to as many as 8 hyo-laryngeal muscles. Stimulation will be coincident with a button press initiation under patient control while eating or at regular intervals for saliva swallows during the day and/or at night. Sensory training will include vibrotactile stimulation to the neck coincident with swallowing under patient control to assist with swallowing while eating or for saliva swallows during the day.

Study population: Persons with chronic (greater than 6 months) dysphagia with risk of aspiration secondary to neurological injury, stroke or chronic neurological disease who currently require enteric feeding or severe dietary restrictions because of risk of aspiration.

Design: A Phase 2 clinical trial with random assignment between two treatment groups with blinded assessment of treatment outcome. Both treatment groups will undergo 2 weeks of device training with a speech pathologist. The implant group will undergo training starting 3 weeks after implantation. They will receive prescriptive training when the levels of muscles stimulation will be established for swallowing. Patients will be trained to press a switch to control the stimulation while they are swallowing. The sensory training group will receive the same amount of training to provide sensory stimulation coincident with attempting to swallow.

Outcome measures: Blinded assessment of risk of aspiration on videofluoroscopy using the NIH Swallowing Safety Scale, and patient administration of the Functional Oral Intake Scale (FOIS) for Dysphagia and the Swallowing Quality of Life Outcomes Tool (SWAL_QOL) prior to treatment and at 3, 6, 9, and 12 months following treatment. Patient administration of the FOIS and SWAL_QOL at 24-months.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Inclusive ages of 18 to 90.
* History of cerebral vascular accident (CVA), brain injury or chronic neurological disease such as Parkinson disease or multiple sclerosis or history of chemoradiation for treatment of head and neck cancer resulting in chronic dysphagia.
* Evidence of pharyngeal phase dysphagia that places the patient at risk for aspiration. Risk for aspiration or frank aspiration will be based on the medical history and evidence from a swallowing study. Absence of aspiration is not cause for exclusion if the risk for aspiration is deemed present due to impaired pharyngeal phase of swallowing as judged by an expert experienced in the evaluation of dysphagia. The patient may demonstrate evidence of aspiration or the risk for aspiration on any consistency, perhaps secondary to pharyngeal retention. Aspiration is defined as passage of food, liquid, or secretions into the trachea below the level of the vocal folds. Impaired pharyngeal phase of swallowing may be evidenced by pharyngeal delay, reduced hyolaryngeal elevation, reduced laryngeal closure, and reduced pharyngeal clearance of the bolus. Signs of pharyngeal delay include temporary pooling of the material in the vallecula with eventual spill over into the pyriform sinuses. Reduced hyolaryngeal elevation will be identified when the larynx is not protected by epiglottal lowering and remains opens to the bolus during a swallow on videoendoscopy. Reduced pharyngeal clearance can be seen during videoendoscopy when the bolus remains in the vallecula and/or pyriform sinuses.
* Other criteria for inclusion for subjects who do not meet the criteria of having aspiration on videofluoroscopy because of the limited number of swallows necessitated by radiation exposure, or who are noncompliant with their NPO status are:

  1. Not all of the bolus can enter the esophagus because of reduced opening of the upper esophageal sphincter, as a result there is pooling of the bolus in the pyriform sinuses which will spill over into the airway.
  2. Many patients who have had dysphagia for several years, have learned to cough up the bolus from the hypopharynx and spit it out, thus preventing aspiration but are continuing to be unable to ingest food or liquid. This is how they manage their accumulation of saliva by spitting in a cup throughout the day. In this way although they cannot swallow they do not aspirate on examination; rather they clear back up any remaining bolus up into their mouths.
  3. Other signs of risk of aspiration are the observation of liquid or food remaining in the pyriform sinuses, a wet gurgling sound during phonation indicating that there is pooling at the vocal folds and coughing when the bolus has already entered the trachea on attempts to swallow.
* Duration of Dysphagia for 6 months or more.
* A score of 2 or greater on the NIH Swallowing Safety Scale.
* Participants may have other health problems such as diabetes mellitus, arteriosclerotic coronary vascular disease and a history of smoking. These will not be cause for automatic exclusion, but will be examined on an individual basis by the otolaryngologist in determining the potential risk and benefit to the individual participant.
* Prior history of tracheostomy is not a cause for exclusion. Patients currently with a tracheostomy will be excluded.
* Restricted oral intake. Patients should demonstrate a current dependence on alternate means of nutrition and hydration (PEG, PEJ); however, PO intake is not cause for exclusion.
* Adequate cognitive skills as demonstrated by a Mini-Mental State Examination (MMSE) score greater than or equal to 23.
* Stable medical status. To determine if a patient has stable medical status prior to admission, the patient will be asked to provide a letter from their physician stating that the patient is medically stable and may participate in the study.

EXCLUSION CRITERIA:

* Subjects with Severe or Very Severe Chronic Obstructive Pulmonary Disorder (COPD). Definition of Severe COPD is an FEV(1)/FVC ratio of less than 70% and an FEV(1) of 30 to less than 50% of predicted. The definition of Very severe COPD is an FEV(1)/FVC ratio of less than 70% and an FEV(1) of less than 30% of predicted. Spirometry will be performed according to the standards of the American Thoracic Society using reference values that include a correction for race.
* HIV positive or immune compromised. This is essential because increased risk of immune reactions to the implantation of a foreign device in patients who are immune compromised. Such patients would be at much greater risk of an infection with implantation of a device. Participation would more likely lead to the need an explanation and a second surgery.
* Patients with a pacemaker, deep brain stimulator or other indwelling electrical device.
* History of rapidly progressive neurodegenerative disorders, such as progressive supranuclear palsy, dementia, peripheral neuropathy, multiple systems atrophy or amyotrophic lateral sclerosis.
* Severe oral phase swallowing deficits, due to loss of tongue control, that prevent bolus retention in the oral cavity.
* No aspiration or risk for aspiration in previous assessment or during preliminary studies.
* An esophageal motility disorder preventing food or liquid from adequately moving through the esophagus into the stomach.
* Pregnant women will be excluded from participation because the study involves radiation exposure.
* Current psychiatric disorder other than depression. Examples of psychiatric disorders to be excluded are: somatoform disorders, conversion disorders, schizophrenia or bipolar disorder.
* Inability to coordinate button press with swallow (as determined during screening).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-07; Primary Completion 2010-09 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Crary MA, Mann GD, Groher ME. Initial psychometric assessment of a functional oral intake scale for dysphagia in stroke patients. Arch Phys Med Rehabil. 2005 Aug;86(8):1516-20. doi: 10.1016/j.apmr.2004.11.049. PMID 16084801
- [Background] McHorney CA, Bricker DE, Kramer AE, Rosenbek JC, Robbins J, Chignell KA, Logemann JA, Clarke C. The SWAL-QOL outcomes tool for oropharyngeal dysphagia in adults: I. Conceptual foundation and item development. Dysphagia. 2000 Summer;15(3):115-21. doi: 10.1007/s004550010012. PMID 10839823
- [Background] Kahrilas PJ, Lin S, Rademaker AW, Logemann JA. Impaired deglutitive airway protection: a videofluoroscopic analysis of severity and mechanism. Gastroenterology. 1997 Nov;113(5):1457-64. doi: 10.1053/gast.1997.v113.pm9352847.
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2006-N-0212.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Vibrotactile: An external vibrotactile device used for swallowing retraining
- Intramuscular: An implanted neurostimulator device used for swallowing retraining
Period: Overall Study
Arm/Group | Vibrotactile | Intramuscular
Started | 4 | 6
Completed | 4 | 4
Not Completed | 0 | 2
Not completed — Death | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vibrotactile | Intramuscular | Total
Number analyzed (Participants) | 4 | 6 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 3
  >=65 years | 3 | 4 | 7
Age Continuous [Mean (Standard Deviation); unit: years] | 70.25 (13.2003) | 61.16 (17.702) | 64.8 (15.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Swallowing Safety for 10 ml of Thin Liquid
Description: Every 3 months swallowing safety was measured using the Swallowing Safety Scale (SSS). The SSS measures 11 swallowing variables including: the presence of residue in the valleculae, laryngeal vestibule, and/or pyriform sinuses, the presence of penetration arising from the oropharynx and/or the hypopharynx, the number of aspiration events arising from the oropharynx and/or the hypopharynx, response to aspiration, degree of esophageal entry, presence of regurgitation, and the presence of >1 swallow per bolus. Scores range from 0 (safe swallowing) to >5 (severely impaired swallowing safety). The maximum score is infinite as the number of occurrences of aspiration is counted in the total score. A higher score on the SSS indicates reduced swallowing safety. Swallows of 10 ml thin liquid, were captured during videofluoroscopy. The SSS was scored from videotaped swallows, by speech pathologists. The raters were blinded to the identity of the patient, group, and time post training.
Time Frame: Baseline and 12-months post-treatment
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Vibrotactile: Patients utilized an external vibrotactile device placed on the thyroid cartilage. Patients were trained to initiate a swallow within 500 ms of stimulation. Stimulation was induced by a patient operated handheld controller. Patients were instructed to perform 60 trials per day.
- Intramuscular: Patients used a surgically implanted intramuscular stimulation device. Patients were trained to initiate a swallow within 500 ms of stimulation. Stimulation was induced by a patient operated handheld controller. Patients were instructed to perform 60 trials per day.
Arm/Group | Vibrotactile | Intramuscular
Number analyzed (Participants) | 4 | 4
units on a scale
  Baseline | 8.417 (0.540) | 7.167 (1.347)
  12-months | 8.250 (3.167) | 7.375 (1.250)

2. Secondary Outcome: Penetration-Aspiration Scale for 10 ml Thin Liquid
Description: Every 3 months swallowing was measured using the Penetration-Aspiration (P/A) Scale. The P/A scale is an 8-point interval scale measuring the depth to which material passes into the airway and the patients cough response. A score of 0 indicates no penetration or aspiration. A score of 8 indicates the presence of aspiration with no cough response. A higher score indicates reduced swallowing safety. Swallows of 10 ml thin liquid, were captured during videofluoroscopy. The P/A Scale was scored by speech pathologists blinded to the identity of the patient, group, and time post training, from videotaped swallows.
Time Frame: Baseline and 12-months post-treatment
Population: intention to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Intramuscular: Patients utilized an implanted neurostimulator device for swallowing. Patients were trained to initiate a swallow within 500 ms of stimulation. Stimulation was induced by a patient operated handheld controller. Patients were instructed to perform 60 trials per day.retraining
Arm/Group | Vibrotactile | Intramuscular
Number analyzed (Participants) | 4 | 4
units on a scale
  Baseline | 5.792 (0.854) | 5.000 (1.700)
  12 months | 5.792 (2.451) | 4.292 (2.266)

3. Secondary Outcome: Penetration-Aspiration Scale for 5 ml Pudding
Description: Every 3 months swallowing was measured using the Penetration-Aspiration (P/A) Scale. The P/A scale is an 8-point interval scale measuring the depth to which material passes into the airway and the patients cough response. A score of 0 indicates no penetration or aspiration. A score of 8 indicates the presence of aspiration with no cough response. A higher score indicates reduced swallowing safety. Swallows of 5 ml pudding, were captured during videofluoroscopy. The P/A Scale was scored by speech pathologists blinded to the identity of the patient, group, and time post training, from videotaped swallows.
Time Frame: Baseline and 12-months post-treatment
Population: intention to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Intramuscular: Patients utilized an implanted neurostimulator device for swallowing retraining. Patients were trained to initiate a swallow within 500 ms of stimulation. Stimulation was induced by a patient operated handheld controller. Patients were instructed to perform 60 trials per day.
Arm/Group | Vibrotactile | Intramuscular
Number analyzed (Participants) | 4 | 4
units on a scale
  Baseline | 1.417 (0.419) | 2.083 (1.067)
  12 months | 2.333 (1.097) | 1.458 (0.417)

4. Primary Outcome: Swallowing Safety for 5 ml of Pudding
Description: as for outcome 1
Time Frame: Baseline and 12-months post-treatment
Population: intention to treat
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Intramuscular: Patients used a surgically implanted intramuscular stimulation device. Patients utilized an external vibrotactile device placed on the thyroid cartilage. Patients were trained to initiate a swallow within 500 ms of stimulation. Stimulation was induced by a patient operated handheld controller. Patients were instructed to perform 60 trials per day.
Arm/Group | Vibrotactile | Intramuscular
Number analyzed (Participants) | 4 | 4
Units on a scale
  Baseline | 6.667 (0.272) | 6.917 (1.664)
  12-months | 6.667 (0.871) | 6.583 (0.441)

5. Secondary Outcome: Functional Oral Intake Scale (FOIS) for Dysphagia
Description: The FOIS was administered at baseline and every 3 months post-treatment during the first year. The FOIS is a 7 point ordinal scale reflecting the functional oral intake of patients. A score of 1 indicates no oral nutrition; a score of 7 indicates all nutrition is taken orally.
Time Frame: Baseline and 12-months post-treatment
Population: intention to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vibrotactile | Intramuscular
Number analyzed (Participants) | 4 | 4
units on a scale
  Baseline | 1.0 (0.0) | 1.0 (0.0)
  12 months | 3.250 (2.630) | 3.0 (.816)

6. Secondary Outcome: Quality of Life Patient Questionnaire
Description: The SWAL-QOL (Swallowing Quality of Life) questionnaire was administered at baseline and every 3 months during the first year. The SWAL-QOL is a 44 item tool that measure 10 quality of life domains, i.e., food selection, burden, mental health, social functioning, fear, eating duration, eating desire, communication, sleep, and fatigue. Scores range from 0 to 100. A lower score indicates greater impairment.
Time Frame: Baseline and 12-months post-treatment
Population: intention to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vibrotactile | Intramuscular
Number analyzed (Participants) | 4 | 4
units on a scale
  Baseline | 55.208 (7.311) | 51.389 (4.598)
  12 months | 68.316 (15.829) | 57.726 (12.281)

ADVERSE EVENTS:
Arm/Group | Vibrotactile | Intramuscular
Serious Adverse Events (participants affected / at risk) | 2/4 | 4/6
Other Adverse Events (participants affected / at risk) | 1/4 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vibrotactile (N=4) | Intramuscular (N=6)
Decreased responsiveness (Nervous system disorders) | 0 (0) | 1 (1)
Neurological symptoms following antibiotic administration (Nervous system disorders) | 1 (1) | 0 (0)
Device malfunction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Nervous system disorders) | 0 (0) | 1 (1)
PEG site problem (Gastrointestinal disorders) | 1 (1) | 0 (0)
Venous occlusion in eye (Eye disorders) | 1 (1) | 0 (0)
Deceased unrelated to study (Nervous system disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vibrotactile (N=4) | Intramuscular (N=6)
Neck irritation at suture site (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Seroma (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Upper Respiratory Infection (Immune system disorders) | 0 (0) | 2 (2)
Complication of aspiration during VSE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Fever (Infections and infestations) | 1 (1) | 0 (0)
Panic Attack (Psychiatric disorders) | 0 (0) | 1 (1)
INS flipped (Investigations) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes